CLINICAL TRIAL: NCT05227404
Title: Evaluation of the Feasibility and Reproducibility of 2 Point-of-Care Tests for SARS-Co-V-2 Antibodies (INSIGHT 017)
Brief Title: Evaluation of Point-of-Care (EPOC) for COVID-19
Acronym: (EPOC)
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00014758
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: COVID-19; SARS CoV 2 Infection
Keywords: COVID-19; SARS COV 2; COVID19 testing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID19 Assays: All participants enrolled will receive 2 point of care assays, and 1 central lab assay
  Interventions: Diagnostic Test: LumiraDX; Diagnostic Test: RightSign; Diagnostic Test: Case Control

INTERVENTIONS:
Diagnostic Test: LumiraDX — Point-of-care test for SARS-CoV-2
Diagnostic Test: RightSign — Point-of-care test for SARS-CoV-2
Diagnostic Test: Case Control — Genscript assay performed on the plasma sample

SUMMARY:
EPOC is designed to examine the feasibility of conducting two point-of-care (POC) tests the LumiraDx SARS-CoV-2 Antibody Test and the RightSign COVID-19 IgG/IgM Rapid Test for SARS-CoV-2 antibodies and compare the reproducibility of these tests to tests run at a central laboratory on specimens obtained from the same study participants at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Informed consent by the patient or the patient's legally authorized representative (LAR) for up to 4 fingersticks for POC testing and a blood draw for stored blood samples.
* SARS-CoV-2 infection, documented by a nucleic acid test (NAT) or equivalent testing within 3 days prior to consent OR documented by NAT or equivalent testing more than 3 days prior to consent AND progressive disease suggestive of ongoing SARS-CoV-2 infection per the responsible investigator. (For non-NAT tests, only those deemed with equivalent specificity to NAT by the protocol team will be allowed. A central list of allowed non-NAT tests is maintained for TICO and that list will also be used for this protocol.)
* Duration of symptoms attributable to COVID-19 ≤ 12 days per the responsible investigator.
* Requiring admission for inpatient hospital acute medical care for clinical manifestations of COVID-19, per the responsible investigator, and NOT for purely public health or quarantine purposes.

Exclusion Criteria:

* Prior receipt of SARS-CoV-2 hIVIG, convalescent plasma from a person who recovered from COVID-19, or SARS-CoV-2 nMAb within 6 months of the blood draws for testing as part of this protocol.
* Disease severity beyond that of stratum 1 in the TICO trial. This includes the following conditions:

  1. stroke
  2. meningitis
  3. encephalitis
  4. myelitis
  5. myocardial infarction
  6. myocarditis
  7. pericarditis
  8. symptomatic congestive heart failure (CHF; New York Heart Association [NYHA] class III-IV)
  9. arterial or deep venous thrombosis or pulmonary embolism
* Current requirement for any of the following:

  1. high-flow supplemental oxygen
  2. non-invasive ventilation
  3. invasive mechanical ventilation
  4. extracorporeal membrane oxygenation
  5. mechanical circulatory support
  6. vasopressor therapy
  7. commencement of renal replacement therapy at this admission (i.e., not patients on chronic renal replacement therapy).
* In the opinion of the responsible investigator, any condition for which, participation would not be in the best interest of the participant or that could limit protocol specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults hospitalized with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reilly C, Mylonakis E, Dewar R, Young B, Nordwall J, Bhagani S, Chia PY, Davis R, Files C, Ginde AA, Hatlen T, Helleberg M, Hayanga A, Jensen TO, Jain MK, Kalomenidis I, Kim K, Lallemand P, Lindegaard B, Menon A, Ognenovska K, Poulakou G, Thorup Roge B, Rogers AJ, Shaw-Saliba K, Sandkovsky U, Trautner BW, Vasudeva SS, Vekstein A, Viens K, Wyncoll J, DuChateau B, Zhang Z, Wu S, Babiker AG, Davey V, Gelijns A, Higgs E, Kan V, Lundgren J, Matthews GV, Lane HC. Evaluation of the Feasibility and Efficacy of Point-of-Care Antibody Tests for Biomarker-Guided Management of Coronavirus Disease 2019. J Infect Dis. 2025 Mar 17;231(3):677-683. doi: 10.1093/infdis/jiae452. PMID 39269490

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COVID19 Assays
Started | 330
Completed | 330
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | COVID19 Assays
Number analyzed (Participants) | 330
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 148
  >=65 years | 182
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153
  Male | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 62
  White | 221
  More than one race | 0
  Unknown or Not Reported | 24

OUTCOME MEASURES:

1. Primary Outcome: Test Results Comparison Between LumiraDx and GenScript
Description: LumiraDx test and GenScript assay are two ways to determine the presence of antibodies to SARS-CoV-2. This measure is a comparison to check agreement between the two tests' results. This is a comparison of the proportion of the positive tests. The comparison is made by looking at the difference of the two proportions obtained by the two tests, so the measure is unitless.
Time Frame: an average of 1 day
Measure: Number (95% Confidence Interval); unit: Unitless
Arm/Group | COVID19 Assays
Number analyzed (Participants) | 330
Unitless | 0.097 [0.059 to 0.135]

2. Primary Outcome: Comparison of Results Obtained by RightSign and GenScript
Description: RightSign test and GenScript assay are two ways to determine the presence of antibodies to SARS-CoV-2. This measure is a comparison to check agreement between the two tests' results. This is a comparison of the proportion of the positive tests. The comparison is made by looking at the difference of the two proportions obtained by the two tests, so the measure is unitless.
Time Frame: an average of 1 day
Measure: Number (95% Confidence Interval); unit: Unitless
Arm/Group | COVID19 Assays
Number analyzed (Participants) | 330
Unitless | -0.038 [-0.074 to -0.001]

3. Secondary Outcome: LumiraDx Valid Test Frequency
Description: The frequency with which the LumiraDx test fails to give an unambiguous result
Time Frame: an average of 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | COVID19 Assays
Number analyzed (Participants) | 330
Participants | 263

4. Secondary Outcome: RightSign Valid Test Frequency
Description: The frequency with wich the RightSign test fails to give an unambiguous result
Time Frame: an average of 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | COVID19 Assays
Number analyzed (Participants) | 330
Participants | 327

ADVERSE EVENTS:
Time Frame: adverse events were not collected
Description: Adverse events were not collected
Arm/Group | COVID19 Assays
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-12-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT05227404/Prot_SAP_ICF_000.pdf